CLINICAL TRIAL: NCT03060304
Title: The Effect of Tamoxifen on Endometrial Thickness and Pregnancy Outcome in Women With Thin Endometrium Undergoing Frozen Thawed Cycle.
Brief Title: The Effect of Tamoxifen on Clinical Outcome in Women With Thin Endometrium Undergoing Frozen Thawed Cycle.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: newivf20170217
Record Dates: First submitted 2017-02-18; First posted 2017-02-23 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Endometrium
Keywords: tamoxifen; thin endometrium; frozen embryo transfer; pregnancy rate
MeSH Terms: interventions — Tamoxifen; Estradiol

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Patients in study group will receive tamoxifen at a daily dose of 40 mg from day 3 to day 8. Follicle diameters are monitored by transvaginal ultrasound and serum levels of E2, P are tested on day 9. If there is a dominant follicle (almost 12 × 12 mm in diameter), endometrial thickness and endometrial pattern, as well as follicular diameters, were monitored daily or every other day till embryo transfer. Serum levels of E2, P are tested on the day before ovulation. If there isn't dominant follicle and intramuscular human menopausal gonadotropin at a dose of 75-150 IU was administered each day after day 12 if there follicle development was poor. The embryo transfer day is decided according embryo development.
  Interventions: Drug: Tamoxifen
- control group (Active Comparator): Patients in control group will receive estradiol valerate at a dose of 3 mg twice per day from day 3. Follicle diameters are monitored by transvaginal ultrasound and serum levels of E2, P are tested on day 9. If endometrial thickness <7mm and E2<100pg/ml, the dose of estradiol valerate can increase or combine other estradiol. Endometrial thickness and endometrial pattern, as well as follicular diameters, were monitored daily or every other day till embryo transfer. Serum levels of E2, P are tested on the day before endometrium transformation. The embryo transfer day is decided according embryo development. Serum levels of E2, P are tested on the day before embryo transfer.
  Interventions: Drug: estradiol valerate

INTERVENTIONS:
Drug: Tamoxifen — Patients in study group will receive tamoxifen at a daily dose of 40 mg from day 3 to day 8.
  Other Names: Tam
  Arms: study group
Drug: estradiol valerate — Patients in control group will receive estradiol valerate at a dose of 3 mg twice per day from day 3.
  Arms: control group

SUMMARY:
Cryopreservation of embryos created during fresh IVF cycles provides a less expensive and time-intensive opportunity for pregnancy. Ideal endometrium thickness is the key point to optimization FET cycle. Researches show that when endometrial thickness is less than 7mm, pregnancy rate dropped significantly. Tamoxifen has been reported to be oestrogenic on the lower genital tract. Several study on intrauterine insemination or ovulation induction suggest that tamoxifen may be a promising alternative for patients with thin endometrium. Based on this ,we want to evaluate the effects of tamoxifen on endometrial thickness and pregnancy outcome in women who failed to develop an adequate endometrial thickness in previous frozen embryo transfer cycle twice or even more times and willing to have another attempt.

DETAILED DESCRIPTION:
Objective: To investigate the effects of tamoxifen on endometrial thickness and pregnancy outcome in women with thin endometrium undergoing frozen thawed cycle.

Study design: This is a single center, randomize control clinical trial. We plan to recruit 100 patients from Mar 2017 to Dec 2019, who failed to develop an adequate endometrial thickness in previous frozen embryo transfer cycle twice or even more times and willing to have another attempt, dividing into two group, one prepare the endometrium through ovulation induction with tamoxifen and progesterone(Study Group), the other is hormone replacement cycle (control group).

Intervention: Study Group will give endometrial preparation with tamoxifen and progesterone, control group will prepared with estrogen and progesterone supplementation.

Main outcome measures: The primary outcome of the study was endometrium thickness and clinical pregnancy rate, the secondary outcomes are cycle duration, cycle cancellation rate, implantation rate, miscarriage rate, live birth rate.

ELIGIBILITY:
Inclusion Criteria:

1. Women age ≥20 years and ≤40 years;
2. patients that have at least 1 high quality blastocysts;
3. patients who are observed endometrial thickness ≤ 7mm in the past natural cycles or hormone replacement cycles repeatedly (twice or even more);
4. patients intends to continue to attempt another frozen embryo transfer cycle.

Exclusion Criteria:

1. patients diagnosed intrauterine adhesions, uterine scarring diverticulum via Hysteroscopy or ultrasonography and have history of uterine cavity operation for the above indication;
2. patients have congenital uterine anomalies such as Gemini, the mediastinum in the uterus and so on.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
endometrium thickness | 1-3 month
  Endometrial thickness was defined as the maximal distance between the echogenic interfaces of the endometrium and the myometrium in the plane of the central longitudinal axis of the uterus.
clinical pregnancy rate | 1-2years
  Clinical pregnancy was considered with the presence of a gestational sac containing yolk sac at transvaginal ultrasonography, including ectopic pregnancy.clinical pregnancy rate is the number of clinical pregnancy patients /the total number of transferred patients in the group.

SECONDARY OUTCOMES:
cycle duration | 1-3 month
  the total time of endometrium preparation
cycle cancellation rate | 1-3 month
  cycle cancellation rate is the number of patients that cancell embryo transfer /the total number of patients in the group.
implantation rate | 1-2 year
  Implantation rate was determined by the number of gestational sacs and the total number of embryos transferred at least 4 weeks after embryo transfer.
miscarriage rate | 1-2 year
  miscarriage rate is the number of patients that find pregnancy loss /the total number of transferred patients in the group.
live birth rate | 1-2 year
  live birth rate is the number of patients that delived /the total number of transferred patients in the group.

CONTACTS AND LOCATIONS:
Overall Officials: Xing Yang, M.D. & Ph.D., Study Director — The Sixth Affiliated Hospital, Sun Yat-sen University